CLINICAL TRIAL: NCT02255279
Title: A Phase 3, Observed-Blind, Randomized, Multi-center Study to Evaluate Safety and Immunogenicity of an Adjuvanted Trivalent Influenza Vaccine in Children 6 to <72 Months of Age in Mexico.
Brief Title: Safety and Immunogenicity of an Adjuvanted Trivalent Influenza Vaccine in Children 6 to <72 Months of Age in Mexico.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V70_50
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aTIV (Experimental): aTIV is a trivalent influenza virus vaccine, adjuvanted with MF59C.
  Interventions: Biological: Adjuvanted Trivalent Influenza Vaccine, 1 dose for non-naive subjects (day 1), two doses for naive subjects (day 1 and day 29)
- TIV (Active Comparator): TIV is trivalent influenza vaccine licensed in Mexico.
  Interventions: Biological: Non-adjuvanted Trivalent Influenza Vaccine, 1 dose for non-naive subjects (day 1), two doses for naive subjects (day 1 and day 29).

INTERVENTIONS:
Biological: Adjuvanted Trivalent Influenza Vaccine, 1 dose for non-naive subjects (day 1), two doses for naive subjects (day 1 and day 29) — A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of aTIV, a trivalent (surface antigen, formaldehyde-inactivated) influenza virus vaccine, adjuvanted with MF59C.1, administered at day 1 (for all subjects) and day 29 (for naïve subjects).
  Arms: aTIV
Biological: Non-adjuvanted Trivalent Influenza Vaccine, 1 dose for non-naive subjects (day 1), two doses for naive subjects (day 1 and day 29). — A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of TIV , an egg-derived trivalent split influenza vaccine licensed in Mexico, administered at day 1 (for all subjects) and day 29 (for naïve subjects)
  Arms: TIV

SUMMARY:
The administration of adjuvanted Trivalent Influenza Vaccine (aTIV) has come to result in a more immunogenic and effective response compared with conventional influenza vaccines in elderly and adults.

The aim of this study is to evaluate safety and immunogenicity of Novartis aTIV in children 6 to <72 months of age, Mexican population, in comparison to Fluzone, a non-adjuvanted trivalent influenza vaccine (TIV).

ELIGIBILITY:
Inclusion Criteria:

* Individuals of >6 months through <72 months of age on the day of informed consent.
* Individuals whose parent(s)/legal guardian(s) have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
* Individuals who can comply with study procedures.
* Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

* Progressive, unstable or uncontrolled clinical conditions.
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
* History of progressive or severe neurologic disorder, seizure disorder or Guillain-Barré syndrome.
* Surgery planned during the study period that in the Investigator's opinion would interfere with the study visits schedule.
* Known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Any fatal prognosis of an underlying medical condition (<12 month life expectancy).
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Abnormal function of the immune system resulting from:

  1. Clinical conditions.
  2. Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 90 days prior to informed consent.
  3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
* Received immunoglobulins or any blood products within 180 days prior to informed consent.
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
* Study personnel as an immediate family or household member.
* Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
* Received any influenza vaccine (licensed or investigational) or with laboratory confirmed influenza within 6 months prior enrollment.
* Received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccines.

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 287 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Mexico (3):
  - 03, Centro Médico Universitario, Colonia Chamilpa, Cuernavaca, Morelos
  - 02, Unidad de Atencion Medica E Investigacion En Salud S.C (Unamis), Mérida, Yucatán
  - 04, Medical Care and Research S.A. de C.V., Mérida, Yucatán

REFERENCES:
- [Derived] Cruz-Valdez A, Valdez-Zapata G, Patel SS, Castelli FV, Garcia MG, Jansen WT, Arora AK, Heijnen E. MF59-adjuvanted influenza vaccine (FLUAD(R)) elicits higher immune responses than a non-adjuvanted influenza vaccine (Fluzone(R)): A randomized, multicenter, Phase III pediatric trial in Mexico. Hum Vaccin Immunother. 2018 Feb 1;14(2):386-395. doi: 10.1080/21645515.2017.1373227. Epub 2018 Jan 3. PMID 28925801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 3 study centers in Mexico.
Pre-assignment Details: All enrolled subjects were included in study.
Groups:
- aTIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of aTIV to be administered.
- TIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of TIV to be administered.
Period: Overall Study
Arm/Group | aTIV (6 Months to < 72 Months) | TIV (6 Months to < 72 Months)
Started | 144 | 143
Completed | 139 | 134
Not Completed | 5 | 9
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aTIV (6 Months to < 72 Months) | TIV (6 Months to < 72 Months) | Total
Number analyzed (Participants) | 144 | 143 | 287
Age, Continuous [Mean (Standard Deviation); unit: Months] | 29.5 (18.2) | 30.1 (19.1) | 29.8 (18.6)
Gender [Count of Participants; unit: Participants]
  FEMALE | 68 | 72 | 140
  MALE | 76 | 71 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Naive Subjects 6 to < 36 Months Old Reporting Solicited Local and Systemic Adverse Events (AEs) From Day 1 to Day 7 Following Each Vaccination.
Description: Number of naive subjects 6 to < 36 months old reporting solicited local and systemic AEs from Day 1 to Day 7 after first vaccination and from Day 29 to Day 35 after second vaccination.
Time Frame: From Day 1 to Day 7 by vaccination
Population: Analysis performed on the Solicited Safety Set.
Measure: Number; unit: Participants
Groups:
- Naive_aTIV (6 to <36 Months): A 0.25 mL (for children 6 to <36 months old) dose of aTIV to be administered.
- Naive_TIV (6 to <36 Months): A 0.25 mL (for children 6 to <36 months old) dose of TIV to be administered.
Arm/Group | Naive_aTIV (6 to <36 Months) | Naive_TIV (6 to <36 Months)
Number analyzed (Participants) | 68 | 69
Participants
  Any Local (Vac-1) | 35 | 20
  Any Local (Vac-2, N= 67,67) | 21 | 15
  Injection site ecchymosis (Vac-1, N= 65,69) | 2 | 2
  Injection site ecchymosis (Vac-2, N= 66,67) | 1 | 1
  Injection site induration (Vac-1, N= 66,69) | 5 | 6
  Injection site induration (Vac-2, N= 66,67) | 3 | 4
  Injection site swelling (Vac-1, N= 65,69) | 8 | 2
  Injection site swelling (Vac-2, N= 66,67) | 2 | 2
  Injection site erythema (Vac-1, N= 64,69) | 9 | 8
  Injection site erythema (Vac-2, N= 66,67) | 7 | 4
  Injection site tenderness (Vac-1, N= 66,69) | 26 | 16
  Injection site tenderness (Vac-1, N= 66,66) | 17 | 13
  Any Systemic (Vac-1) | 34 | 27
  Any Systemic (Vac-2, N=67,67) | 27 | 22
  Body Temperature (>=40°C) (Vac-1, N= 67,68) | 0 | 0
  Body Temperature (>=40°C) (Vac-2, N= 67,67) | 0 | 0
  Fever (Vac-1) | 7 | 5
  Fever (Vac-2, N= 67,67) | 7 | 2
  Change in eating habits (Vac-1, N= 67,69) | 14 | 4
  Change in eating habits (Vac-2, N= 66,67) | 11 | 7
  Diarrhea (Vac-1, N= 67,69) | 15 | 15
  Diarrhea (Vac-2, N= 66,67) | 11 | 11
  Irritability (Vac-1, N= 67,69) | 18 | 13
  Irritability (Vac-2, N= 66,67) | 17 | 9
  Persistent Crying (Vac-1, N= 67,69) | 15 | 11
  Persistent Crying (Vac-2, N= 66,67) | 11 | 9
  Sleepiness (Vac-1, N= 67,68) | 10 | 11
  Sleepiness (Vac-2, N= 65,67) | 8 | 9
  Vomiting (Vac-1, N= 67,68) | 5 | 4
  Vomiting (Vac-2, N= 65,67) | 2 | 2
  Prevention of Pain and or Fever (Vac-1, N= 67,67) | 2 | 2
  Prevention of Pain and or Fever (Vac-2, N= 64,67) | 3 | 2
  Treatment of Pain and or Fever (Vac-1, N= 67,67) | 9 | 7
  Treatment of Pain and or Fever (Vac-1, N= 66,67) | 10 | 2

2. Primary Outcome: Number of Non-naive Subjects 6 to < 36 Months Old Reporting Solicited Local and Systemic AEs From Day 1 to Day 7 After Vaccination.
Description: Number of non-naive subjects 6 to < 36 months old reporting solicited local and systemic AEs from Day 1 to Day 7 after vaccination.
Time Frame: From Day 1 to Day 7
Population: Analysis performed on the Solicited Safety Set.
Measure: Number; unit: Participants
Groups:
- Non-naive_aTIV (6 to <36 Months): A 0.25 mL (for children 6 to <36 months old) dose of aTIV to be administered.
- Non-naive_TIV (6 to <36 Months): A 0.25 mL (for children 6 to <36 months old) dose of TIV to be administered.
Arm/Group | Non-naive_aTIV (6 to <36 Months) | Non-naive_TIV (6 to <36 Months)
Number analyzed (Participants) | 22 | 22
Participants
  Any Local | 10 | 7
  Injection site ecchymosis | 0 | 1
  Injection site induration | 2 | 0
  Injection site swelling | 1 | 1
  Injection site erythema | 2 | 4
  Injection site tenderness (N= 22,21) | 9 | 4
  Any Systemic | 9 | 7
  Body Temperature (>= 40.0°C) | 0 | 0
  Fever | 6 | 1
  Change in eating habits | 4 | 3
  Diarrhea | 3 | 6
  Irritability | 4 | 3
  Persistent Crying | 1 | 1
  Sleepiness | 2 | 0
  Vomiting (N= 21,21) | 1 | 1
  Prevention of Pain and or Fever (N= 21,22) | 0 | 0
  Treatment of Pain and or Fever (N= 21,22) | 2 | 1

3. Primary Outcome: Number of Naive Subjects ≥ 36 Months to < 72 Months Old Reporting Solicited Local and Systemic AEs From Day 1 to Day 7 Following Each Vaccination.
Description: Number of naive subjects ≥ 36 months to < 72 months old reporting solicited local and systemic AEs from Day 1 to Day 7 after first vaccination and from Day 29 to Day 35 after second vaccination.
Time Frame: From Day 1 to Day 7 by vaccination
Population: Analysis performed on the Solicited Safety Set.
Measure: Number; unit: Participants
Groups:
- Naive_aTIV (≥36 Months to < 72 Months): A 0.5 mL (for children ≥36 months to < 72 months old) dose of aTIV to be administered.
- Naive_TIV (≥36 Months to < 72 Months): A 0.5 mL (for children ≥36 months to < 72 months old) dose of TIV to be administered.
Arm/Group | Naive_aTIV (≥36 Months to < 72 Months) | Naive_TIV (≥36 Months to < 72 Months)
Number analyzed (Participants) | 6 | 4
Participants
  Any Local (Vac-1) | 5 | 2
  Any Local (Vac-2, N= 6,3) | 4 | 2
  Injection site ecchymosis (Vac-1) | 0 | 0
  Injection site ecchymosis (Vac-2, N= 6,3) | 0 | 0
  Injection site induration (Vac-1) | 2 | 1
  Injection site induration (Vac-2, N= 6,3) | 2 | 0
  Injection site swelling (Vac-1) | 2 | 0
  Injection site swelling (Vac-2, N= 6,3) | 0 | 0
  Injection site erythema (Vac-1) | 1 | 0
  Injection site erythema (Vac-2, N= 6,3) | 0 | 0
  Injection site pain (Vac-1) | 3 | 2
  Injection site pain (Vac-2, N= 6,3) | 3 | 2
  Any Systemic (Vac-1) | 3 | 1
  Any Systemic (Vac-2, N= 6,3) | 2 | 0
  Fatigue (Vac-1) | 1 | 1
  Fatigue (Vac-2, N= 6,3) | 2 | 0
  Myalgia (Vac-1) | 2 | 0
  Myalgia (Vac-2, N= 6,3) | 1 | 0
  Arthralgia (Vac-1) | 0 | 0
  Arthralgia (Vac-2, N= 6,2) | 0 | 0
  Headache (Vac-1) | 1 | 1
  Headache (Vac-2, N= 6,2) | 1 | 0
  Body Temperature (>= 40.0°C) (Vac-1) | 0 | 0
  Body Temperature (>= 40.0°C) (Vac-2, N= 6,3) | 0 | 0
  Fever (Vac-1) | 2 | 0
  Fever (Vac-2, N= 6,3) | 1 | 0
  Chills (Vac-1) | 0 | 0
  Chills (Vac-2, N= 6,3) | 0 | 0
  Change in Eating Habits (Vac-1, N= 5,4) | 2 | 0
  Change in Eating Habits (Vac-2, N= 6,3) | 0 | 0
  Diarrhea (Vac-1) | 0 | 0
  Diarrhea (Vac-2, N= 6,3) | 0 | 0
  Vomiting (Vac-1) | 0 | 0
  Vomiting (Vac-2, N= 6,3) | 0 | 0
  Prevention of Pain and or Fever (Vac-1, N= 6,2) | 1 | 0
  Prevention of Pain and or Fever (Vac-2, N= 4,2) | 0 | 0
  Treatment of Pain and or Fever (Vac-1, N= 6,2) | 0 | 0
  Treatment of Pain and or Fever (Vac-2, N= 5,2) | 0 | 0

4. Primary Outcome: Number of Non-naive Subjects ≥36 Months to < 72 Months Old Reporting Solicited Local and Systemic AEs From Day 1 to Day 7 Following Each Vaccination.
Description: Number of non-naive subjects ≥36 months to < 72 months old reporting solicited local and systemic AEs from Day 1 to Day 7 after vaccination.
Time Frame: From Day 1 to Day 7
Population: Analysis performed on the Solicited Safety Set.
Measure: Number; unit: Participants
Groups:
- Non-naive_aTIV (≥36 Months to < 72 Months): A 0.5 mL (for children ≥36 months to < 72 months old) dose of aTIV to be administered.
- Non-naive_TIV (≥36 Months to < 72 Months): A 0.5 mL (for children ≥36 months to < 72 months old) dose of TIV to be administered.
Arm/Group | Non-naive_aTIV (≥36 Months to < 72 Months) | Non-naive_TIV (≥36 Months to < 72 Months)
Number analyzed (Participants) | 44 | 41
Participants
  Any Local | 17 | 20
  Injection site ecchymosis | 2 | 1
  Injection site induration | 6 | 3
  Injection site swelling | 4 | 3
  Injection site erythema (N= 43,40) | 6 | 7
  Injection site pain (N= 44,40) | 14 | 16
  Injection site tenderness | 0 | 0
  Any Systemic | 15 | 7
  Fatigue (N= 44,40) | 6 | 2
  Myalgia (N= 44,40) | 7 | 0
  Arthralgia (N= 44,40) | 4 | 0
  Headache (N= 44,40) | 3 | 2
  Body Temperature (>= 40.0°C) (N= 44,40) | 0 | 0
  Fever | 2 | 1
  Chills (N= 44,40) | 2 | 0
  Change in eating habits (N= 44,39) | 8 | 3
  Diarrhea (N= 44,39) | 4 | 3
  Vomiting (N= 44,40) | 2 | 1
  Prevention of Pain and or Fever (N= 42,40) | 0 | 0
  Treatment of Pain and or Fever (N=42,40) | 5 | 0

5. Primary Outcome: Number of Naive Subjects Aged 6 to < 72 Months Reporting All Unsolicited AEs From Day 1 to Day 50.
Description: Number of naive subjects aged 6 to < 72 months reporting all unsolicited AEs, medically attended AEs, AE leading to study withdrawal and serious AEs (SAEs) from Day 1 to Day 50.
Time Frame: From Day 1 to Day 50
Population: Analysis performed on the Unsolicited Safety Set.
Measure: Number; unit: Participants
Groups:
- Naive_aTIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of aTIV to be administered.
- Naive_TIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of TIV to be administered.
Arm/Group | Naive_aTIV (6 Months to < 72 Months) | Naive_TIV (6 Months to < 72 Months)
Number analyzed (Participants) | 74 | 73
Participants
  Any AE | 33 | 28
  At least Possibly related AE | 4 | 4
  SAE | 0 | 0
  At least possibly related SAE | 0 | 0
  AE leading to study withdrawal | 0 | 0
  Medically attended AE | 26 | 25
  Death | 0 | 0

6. Primary Outcome: Number of Non-naive Subjects Aged 6 to < 72 Months Reporting All Unsolicited AEs From Day 1 to Day 22
Description: Number of non-naive subjects aged 6 to < 72 months reporting all unsolicited AEs, medically attended AEs, AE leading to study withdrawal and SAEs from Day 1 to Day 22.
Time Frame: From Day 1 to Day 22
Population: Analysis performed on the Unsolicited Safety Set.
Measure: Number; unit: Participants
Groups:
- Non naive_aTIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of aTIV to be administered.
- Non naive_TIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of TIV to be administered.
Arm/Group | Non naive_aTIV (6 Months to < 72 Months) | Non naive_TIV (6 Months to < 72 Months)
Number analyzed (Participants) | 66 | 64
Participants
  Any AE | 9 | 6
  At least Possibly related AE | 2 | 0
  SAE | 0 | 0
  At least possibly related SAE | 0 | 0
  AE leading to study withdrawal | 0 | 0
  Medically attended AE | 3 | 4
  Death | 0 | 0

7. Primary Outcome: Geometric Mean Titers (GMTs), in All Three Homologous Virus Strains in Subjects 6 to < 72 Months of Age.
Description: Antibody response was assessed in terms of GMTs in all three homologous virus strains, 21 days after last immunization, in subjects 6 to <72 months of age.
  The study is considered a success if the 21 days after last immunization GMT ratios of aTIV relative to TIV demonstrate as non-inferior with the lower limit (LL) of the two sided 95% confidence interval (CI) above 0.67 (-0.176 on log10 scale) for each vaccine strain (Center for Biologics Evaluation and Research {CBER} Guideline on Seasonal Vaccines May 2007).
Time Frame: Day 1 and Day 22 (vaccine non-naïve subjects) or Day 50 (vaccine naïve subjects) post vaccination
Population: Analysis performed on the Per Protocol Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | aTIV (6 Months to < 72 Months) | TIV (6 Months to < 72 Months)
Number analyzed (Participants) | 114 | 112
Titers
  A/H1N1 (Day 1) (N= 113,112) | 14 [11 to 19] | 15 [11 to 20]
  A/H1N1 (Day 22 or Day 50) | 675 [536 to 849] | 166 [132 to 208]
  A/H3N2 (Day 1) | 59 [40 to 86] | 55 [38 to 81]
  A/H3N2 (Day 22 or Day 50) | 1280 [1077 to 1521] | 495 [417 to 588]
  B (Day 1) | 7.47 [6.41 to 8.71] | 6.92 [5.95 to 8.06]
  B (Day 22 or Day 50) | 76 [61 to 93] | 16 [13 to 20]
Statistical Analysis 1: Comparison: aTIV (6 Months to < 72 Months) vs TIV (6 Months to < 72 Months); Geometric mean titers (GMTs), in H1N1 strain of all the tree strains in Subjects 6 to < 72 months of Age; Test type: Non-Inferiority or Equivalence — Hypothesis: Demonstrate non-inferiority (NI) of aTIV to TIV: H0 : μAi - μBi ≤ -0.176 (Null) H1 : μAi - μBi >-0.176 (alternative) (i= H1N1, H3N2, B) μA and μB are means of log10-transformed titers 21 days after last vaccination of the aTIV & TIV vaccine groups respectively. NI is claimed if LL of 95% CI for GMT ratios is >0.67. Significance level is α = 2.5% (1-sided), which needs no further adjustment for multiplicity as to reach NI, above hypothesis needs to be rejected for all 3 strains; ANCOVA; Ratio of GMTs = 4.06, 95% CI 2-sided [3.00 to 5.51]
Statistical Analysis 2: Comparison: aTIV (6 Months to < 72 Months) vs TIV (6 Months to < 72 Months); Geometric mean titers (GMTs), in H3N2 strain of all three homologous virus strains in Subjects 6 to < 72 months of Age; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 7, analysis 1]; ANCOVA; Ratio of GMTs = 2.58, 95% CI 2-sided [2.05 to 3.25]
Statistical Analysis 3: Comparison: aTIV (6 Months to < 72 Months) vs TIV (6 Months to < 72 Months); Geometric mean titers (GMTs), in B strain of all three homologous virus strains in Subjects 6 to < 72 months of Age; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 7, analysis 1]; ANCOVA; Ratio of GMTs = 4.67, 95% CI 2-sided [3.52 to 6.20]

8. Secondary Outcome: Percentages of Subjects Achieving Seroconversion in Hemagglutination Inhibition (HI) Titers and Vaccine Group Differences at Day 1 and 21 Days After Last Vaccination With aTIV or TIV in Naive and Non-naive Subjects.
Description: Percentages of subjects with seroconversion in all three homologous virus strains, 21 days after last immunization, in subjects 6 to <72 months of age, defined as: HI ≥ 40 subject with a pre-vaccination HI titer <10; a minimum 4-fold increase HI titer for subjects with a prevaccination HI titer ≥10, on Day 22 (non-naive subjects) or Day 50 (naive subjects), as applicable.
Time Frame: Day 1 and Day 22 (vaccine non-naive subjects) or Day 50 (vaccine naive subjects) post vaccination
Population: Analysis performed on the Per Protocol Set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | aTIV (6 Months to < 72 Months) | TIV (6 Months to < 72 Months)
Number analyzed (Participants) | 114 | 112
Percentages of subjects
  H1N1 strain (N= 113,112) | 90 [83.2 to 95] | 75 [65.9 to 82.7]
  H3N2 strain | 77 [68.4 to 84.5] | 67 [57.4 to 75.6]
  B strain | 78 [69.4 to 85.3] | 22 [15 to 31.2]
Statistical Analysis 1: Comparison: aTIV (6 Months to < 72 Months) vs TIV (6 Months to < 72 Months); Percentage of subjects achieving seroconversion in H1N1 strain after last vaccination with aTIV or TIV in naïve and non-naive subjects; Test type: Non-Inferiority or Equivalence — The following hypotheses should be tested to demonstrate non-inferiority of aTIV to TIV: H0i: πi1 > πi2-0.1 vs. H1i: πi1 > πi2- 0.1 where H0i and H1i represent the null and the alternative hypothesis (respectively) of the non- inferiority objective and πi1 and πi2 represent the seroresponse rates 21 days after last immunization of the aTIV and TIV vaccine groups respectively in the i-th strain (H1N1, H3N2, B). The non-inferiority criterion is -0.1 (i.e., -10%); Loglinear model; Binary data were analyzed using loglinear models with a qualitative factor for vaccine group (αik, i = A, B) and center (δlk, k=1); Vaccine Group Differences = 17, 95% CI 2-sided [8.1 to 26.3]
Statistical Analysis 2: Comparison: aTIV (6 Months to < 72 Months) vs TIV (6 Months to < 72 Months); Percentage of subjects achieving seroconversion in H3N2 strain after last vaccination with aTIV or TIV in naive and non-naive subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; Loglinear model; [statistical method as in outcome 8, analysis 1]; Vaccine Group Differences = 10, 95% CI 2-sided [-1.8 to 21]
Statistical Analysis 3: Comparison: aTIV (6 Months to < 72 Months) vs TIV (6 Months to < 72 Months); Percentage of subjects achieving seroconversion in B strains after last vaccination with aTIV or TIV in naïve and non naive subjects; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; Loglinear model; [statistical method as in outcome 8, analysis 1]; Vaccine Group Differences = 58, 95% CI 2-sided [47.5 to 68.5]

9. Secondary Outcome: Geometric Mean Ratios (GMRs) of HI and Vaccine Group Differences at Day 1 and 21 Days After Last Vaccination With aTIV or TIV in Naive and Non-naive Subjects.
Description: GMRs of HI, day 22/day 1 (non-naive subjects) or day 50/day 1 (naive subjects) in all three homologous virus strains, 21 days after last immunization, in subjects 6 to <72 months of age. As the non-inferiority of aTIV to TIV has been established, GMT ratio of aTIV relative to TIV in all three homologous virus strains, 21 days after last immunization in subjects 6 to <72 months of age was evaluated using margins greater than the non-inferiority cut-off of 0.67.
Time Frame: Day 1 and Day 22 (vaccine non-naive subjects) or Day 50 (vaccine naive subjects) post vaccination
Population: Analysis performed on the Per Protocol Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | aTIV (6 Months to < 72 Months) | TIV (6 Months to < 72 Months)
Number analyzed (Participants) | 114 | 112
Ratios
  H1N1 strain (N=113,112) | 46 [34 to 62] | 11 [8.12 to 15]
  H3N2 strain | 21 [16 to 28] | 8.39 [6.26 to 11]
  B strain | 10 [8.25 to 13] | 2.30 [1.84 to 2.87]

10. Secondary Outcome: Percentages of Subjects With a HI Titer ≥ 40, ≥110 and ≥330 and Vaccine Group Differences at Day 1 and 21 Days After Last Vaccination With aTIV or TIV in Naive and Non-naive Subjects.
Description: Percentage of subjects with a HI titer ≥ 40, ≥110 and ≥330 on Day 1, Day 22 (non naïve subjects) or Day 50 (naïve subjects), in all three homologous virus strains, 21 days after last immunization, in subjects 6 to <72 months of age.
Time Frame: Day 1 and Day 22 (vaccine non-naive subjects) or Day 50 (vaccine naive subjects) post vaccination
Population: Analysis performed on the Per Protocol Set.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | aTIV (6 Months to < 72 Months) | TIV (6 Months to < 72 Months)
Number analyzed (Participants) | 114 | 112
Percentage of subjects
  H1N1 strain (HI titer ≥ 40, Day 1) (N=113,112) | 32 [23.4 to 41.3] | 33 [24.4 to 42.6]
  H1N1 strain (HI titer ≥ 40, Day 22 or Day 50) | 99 [95.2 to 99.98] | 88 [81 to 93.7]
  H1N1 strain (HI titer ≥ 110, Day 1) (N=113,112) | 19 [11.9 to 27] | 20 [12.7 to 28.2]
  H1N1 strain (HI titer ≥ 110, Day 22 or Day 50) | 96 [90.1 to 98.6] | 68 [58.4 to 76.4]
  H1N1 strain (HI titer ≥ 330, Day 1) | 4 [1.5 to 10] | 7 [3.1 to 13.6]
  H1N1 strain (HI titer ≥ 330, Day 22 or Day 50) | 78 [69.4 to 85.3] | 37 [27.7 to 46.2]
  H3N2 strain (HI titer ≥ 40, Day 1) | 56 [46.5 to 65.4] | 58 [48.3 to 67.3]
  H3N2 strain (HI titer ≥ 40, Day 22 or Day 50) | 100 [96.8 to 100] | 97 [92.4 to 99.4]
  H3N2 strain (HI titer ≥ 110, Day 1) | 44 [34.6 to 53.5] | 44 [34.4 to 53.4]
  H3N2 strain (HI titer ≥ 110, Day 22 or Day 50) | 99 [95.2 to 99.98] | 84 [75.8 to 90.2]
  H3N2 strain (HI titer ≥ 330, Day 1) | 33 [24.8 to 42.8] | 30 [22 to 39.8]
  H3N2 strain (HI titer ≥ 330, Day 22 or Day 50) | 86 [78.2 to 91.8] | 61 [51 to 69.8]
  B strain (HI titer ≥ 40, Day 1) | 9 [4.3 to 15.5] | 9 [4.4 to 15.8]
  B strain (HI titer ≥ 40, Day 22 or Day 50) | 84 [76.2 to 90.4] | 32 [23.6 to 41.6]
  B strain (HI titer ≥ 110, Day 1) | 2 [0.21 to 6.2] | 1 [0.02 to 4.9]
  B strain (HI titer ≥ 110, Day 22 or Day 50) | 43 [33.7 to 52.6] | 6 [2.5 to 12.5]
  B strain (HI titer ≥ 330, Day 1) | 0 [0 to 3.2] | 0 [0 to 3.2]
  B strain (HI titer ≥ 330, Day 22 or Day 50) | 8 [3.7 to 14.5] | 0 [0 to 3.2]

ADVERSE EVENTS:
Time Frame: Throughout the study; Day 1 - Day 50 (naive subjects) and Day 1 - Day 22 (non-naive subjects).
Description: Solicited AEs were collected by the subject parent(s)/legal guardian(s) for 7 days from the day of vaccination/s (Day 1 & Day 29 for naive; Day 1 for non-naive). Unsolicited AEs were collected from Day 1 to Day 50 for naive, from Day 1 to Day 22 for non-naive.
  All AEs were monitored until resolution or the investigator assesses them as stable.
Groups:
- Naive_aTIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of aTIV to be administered (Naive).
- Naive_TIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of TIV to be administered (Naive).
  Enrolled subjects- 79 Exposed subjects- 78 Reason for discrepancy- Before vaccination one subject was withdrawn from study because of the suspected egg allergy.
- Non-naive_aTIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of aTIV to be administered (Non-naive).
- Non-naive_TIV (6 Months to < 72 Months): A 0.25 mL (for children 6 to <36 months old) and 0.5 mL (for children ≥36 months to < 72 months old) dose of TIV to be administered (Non-naive).
Arm/Group | Naive_aTIV (6 Months to < 72 Months) | Naive_TIV (6 Months to < 72 Months) | Non-naive_aTIV (6 Months to < 72 Months) | Non-naive_TIV (6 Months to < 72 Months)
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/78 | 0/67 | 0/64
Other Adverse Events (participants affected / at risk) | 58/77 | 52/78 | 35/67 | 31/64
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naive_aTIV (6 Months to < 72 Months) (N=77) | Naive_TIV (6 Months to < 72 Months) (N=78) | Non-naive_aTIV (6 Months to < 72 Months) (N=67) | Non-naive_TIV (6 Months to < 72 Months) (N=64)
Diarrhoea (Gastrointestinal disorders) | 22 | 21 | 7 | 9
Vomiting (Gastrointestinal disorders) | 7 | 6 | 4 | 2
Crying (General disorders) | 20 | 15 | 1 | 1
Fatigue (General disorders) | 3 | 1 | 6 | 2
Injection site erythema (General disorders) | 13 | 11 | 8 | 11
Injection site induration (General disorders) | 10 | 10 | 8 | 3
Injection site pain (General disorders) | 33 | 25 | 23 | 20
Injection site swelling (General disorders) | 12 | 2 | 5 | 4
Pyrexia (General disorders) | 16 | 11 | 9 | 2
Conjunctivitis (Infections and infestations) | 0 | 4 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 16 | 8 | 2 | 2
Pharyngitis (Infections and infestations) | 6 | 10 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 7 | 0
Somnolence (Nervous system disorders) | 16 | 14 | 2 | 0
Eating disorder (Psychiatric disorders) | 20 | 9 | 12 | 6
Irritability (Psychiatric disorders) | 25 | 17 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.